CLINICAL TRIAL: NCT05227417
Title: A Mobile Phone Short Message Service Intervention to Increase Retention in HIV Care Among HIV-Positive Men Who Have Sex With Men in Peru (WELTEL PERU)
Brief Title: A Mobile Phone SMS Intervention to Increase Retention in HIV Care Among HIV-Positive MSM in Peru (WELTEL PERU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WelTel Peru; 1K43TW011428 (NIH)
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-05

CONDITIONS: Retention in Care; Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 2 parallel arms: intervention and control.
Who Masked: Care Provider
Masking Description: The recruiter will be masked to the group assignment. Participants will be randomized after signing the consent form. Because of the nature of the study, healthcare providers and participants will not be masked to group assignment during the delivery of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): SMS-based intervention delivered with a web-based system, which will include weekly health check-ins, appointment reminders all delivered via SMS (text messages).
  Interventions: Behavioral: SMS
- Control (No Intervention): Standard of care: Those who test positive in both tests receive post-test counseling, including emotional support, and are linked to a facility for antiretroviral (ART) initiation, ideally within one week. During the 1st medical appointment after diagnosis, lab tests are requested including CD4 and viral load. In most cases, ART initiation occurs at the second medical appointment when safety lab results are available. Currently, it is not mandatory to have CD4/VL results available to start ART. It is recommended that patients have CD4 counts and viral load assessed twice during the first year. A one-month supply of ART is provided initially. If clients are adherent, ART is dispensed every 3 months by nurses who also assess adherence. Standard follow-up is performed by nurses when clients visit the center for their appointments.

INTERVENTIONS:
Behavioral: SMS — Weekly text messages that will be sent automatically by a web-based system to participants' cell-phones. Participants will be able to respond and messages will reach the system. The health providers will be in charge to respond (from the web system) to participants who reply asking for support or any other request.
  Arms: Intervention

SUMMARY:
We will use a web-based system in order to deliver a text messaging-based intervention and assess the efficacy to increase retention in HIV care among HIV+ gay men in Peru.

DETAILED DESCRIPTION:
We will determine the efficacy of the SMS-based intervention delivered through a web-based system for increasing retention in HIV care when compared with standard-of-care. We will perform a randomized controlled trial. The main outcome will be retention in HIV care within 1 year after enrollment. Participants will be categorized as retained if they attend three medical appointments for HIV care that are separated by 90 days within a one-year period (at the study clinic). Otherwise they will be classified as not retained. The follow-up period will last 6 months. We will identify and recruit 208 HIV+ MSM over a 12-month period at the research site. Healthcare providers at the clinic will be trained to assess eligibility and obtain consent for this study. After enrollment, the recruiter, who will be masked to the group assignment, will obtain consent and give instructions to all participants on how they should interact if they start receiving SMS (text messages). Participants will be randomized after signing the consent form. They will be assigned a study ID and randomly assigned to the intervention or control arm, 1:1 ratio using computer generated random numbers. Allocations will be sealed in individual, sequentially numbered opaque envelopes. The trained providers in charge of delivering the intervention will be informed when a new participant in the intervention arm is enrolled. Because of the nature of the study, healthcare providers and participants will not be masked to group assignment during the delivery of the intervention. Participants allocated to the intervention arm will have their phones registered into the platform.

ELIGIBILITY:
Inclusion Criteria:

1. Be men who have sex with men;
2. Be 18 years or older;
3. Have been diagnosed HIV positive;
4. Own a cell phone which can send and receive text messages;
5. Reside in Lima, Peru;

Exclusion Criteria:

1) Be enrolled in an interventional trial using text messages.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-05-12 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Retention in HIV care | 1 year
  The main outcome will be retention in HIV care within 1 year after enrollment. Participants will be categorized as retained if they attend three medical appointments for HIV care that are separated by 90 days within a one-year period (at the study clinic). Otherwise they will be classified as not retained.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Cayetano Heredia, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT05227417/Prot_SAP_ICF_000.pdf